CLINICAL TRIAL: NCT04750590
Title: Relationship Between Methods of Bladder Tumor Extraction and Local Recurrence Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERBT -MORC20
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Morcellation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- en bloc resection group (Experimental): Patients scheduled for laser en bloc tumor resection with subsequent morcellation of exophytic part of the tumor
  Interventions: Procedure: en bloc resection, morcellation
- piecemeal resection group (Experimental): Patients scheduled for piecemeal bladder tumor TUR with subsequent removing of tissue using the instrument loop or Janet's syringe.
  Interventions: Procedure: piecemeal resection, tissue removal by loop

INTERVENTIONS:
Procedure: en bloc resection, morcellation — Laser en bloc resection with subsequent tumor morcellation will be performed. This tissue will be sent for histology in order to estimate the histological subtype and differentiation grade. Next stage laser resection of the tumor basis will be performed with subsequent histology to determine the depth of invasion and the status of surgical margin.
  Arms: en bloc resection group
Procedure: piecemeal resection, tissue removal by loop — Tumor piecemeal resection will be performed with electric loop. Then fragments of the tumor will be removed by the loop or Janet's syringe. Fragments from the base of the tumor will be sent separately in order to assess which stage the tumor is at and its surgical margin status.
  Arms: piecemeal resection group

SUMMARY:
According to clinical guidelines, endoscopic surgery (mono- or bipolar TURBT, laser resection, en bloc resection) is a standard treatment option for patients with primary non-muscle invasive bladder cancer (NMIBC) (excluding carcinoma in-situ). However, more than half of patients will experience local recurrence after surgery. It is believed that one of the main causes for this local recurrence is the reimplantation of tumor cells during endoscopic surgery. It is crucial to limit contact between the resected tumor and the bladder wall during the operation and to extract the specimen as quickly as possible. In the case of a small tumor, the surgeon can immediately remove it using an endoscopic instrument. There are a number of methods available for removing large tumors, but it is not yet clear which one is most optimal. Therefore, comparing the oncological results from evacuating bladder tumors using various methods is very timely.

Based on the previously mentioned studies, the investigators assume that the rate of bladder cancer relapse out site of the resection area would be lower in the morcellation group compared with piecemeal resection of the tumor. In order to prove this, the investigators plan to conduct a randomized study comparing the relapse rate in these two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for endoscopic bladder tumor removal
2. Non-muscle invasive bladder cancer on contrast-enhanced MRI or CT (stage cT1N0M0 and lower)
3. Diameter of tumor >3cm

Exclusion Criteria:

1. Patient refused to participate in the trial
2. Multiple (more than 2) bladder tumors
3. Previous cold-cup biopsy or any other surgery for bladder tumor
4. Muscle-invasive bladder cancer on postoperative histological evaluation
5. Other malignant/benign tumors of the bladder (non-urothelial cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-04-11 (Estimated); Study Completion 2022-06-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | 3 months
  Absence of the tumor in the bladder during the follow-up cystoscopy

SECONDARY OUTCOMES:
Relapse-free rate in-site of previous surgery | 3 months
  Absence of the tumor in the place of resection of the bladder wall during the follow-up cystoscopy
Relapse-free rate out-site of previous surgery | 3 months
  Absence of the tumor out of the place of resection of the bladder wall during the follow-up cystoscopy
Duration of surgery | Intraoperatively
  Time frame from the beginning of the procedure till the end of the procedure
Adverse events | 3 months
  Adverse events according to the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Enikeev, M.D., Principal Investigator — Sechenov University
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No